| Clinical Study Title | A prospective, single-site, open-label, pharmacokinetic study of intermittent intraperitoneal vancomycin in adult subjects receiving automated peritoneal dialysis (APD) |
|---|---|
| <b>Clinical Study Site</b> | Thomas Jefferson University, Philadelphia, PA |
| Principal | Walter K. Kraft, M.D. |
| Investigator | Department of Pharmacology & Experimental Therapeutics |
| | Thomas Jefferson University Hospital |
| | 132 S. 10 <sup>th</sup> Street, 1170 Main Building |
| | Philadelphia, PA 19107 |
| Co-Investigators Edwin Lam, Pharm.D. | |
| | Jingjing Zhang, M.D., Ph.D. |
| <b>Protocol Date</b> | 13 December 2017 |
| NCT | NCT03685747 |

### **Version History**

| Version | Date | Change History |
|---|---|---|
| 1.0 | 13 December 2017 | Concept Protocol |
| 1.1 | 04 January 2018 | Draft Protocol |
| 2.0 | 03 February 2018 | Protocol |
| 3.0 | 14 September 2018 | Protocol Revision |
| 4.0 | 15 January 2019 | Amendment- Clarification of post-study follow-up, addition of serum creatinine analysis, and clarification on sampling points |

### **Abbreviations**

| APD | Automated Peritoneal Dialysis |
|------|-------------------------------------------|
| AUC | Area Under Concentration-Time Curve |
| CAPD | Continuous Ambulatory Peritoneal Dialysis |
| ESRD | End Stage Renal Disease |
| MIC | Minimum Inhibitory Concentration |
| NCA | Non-Compartmental Analysis |
| PET | Peritoneal Equilibration Test |
| PK | Pharmacokinetics |
| PD | Peritoneal Dialysis |

| 12<br>13 | Table | of Contents | |
|----------|----------|------------------------------------------|----|
| 14 | | | |
| 15 | 1. INTRO | DDUCTION | 3 |
| 16 | 2. STUDY | Y OBJECTIVES | 5 |
| 17 | 2.1 | Primary Objective | 5 |
| 18 | 2.2 | Secondary Objectives | 5 |
| 19 | 3. STUDY | Y DESIGN | 5 |
| 20 | 3.1 | Overview and Design | 5 |
| 21 | 3.2 | Schedule & Procedures | 7 |
| 22 | 4. STUDY | Y POPULATION | 10 |
| 23 | 4.1 | Inclusion Criteria | 10 |
| 24 | 4.2 | Exclusion Criteria | 10 |
| 25 | 5. STUDY | Y ENDPOINTS | 10 |
| 26 | 5.1 Pri | imary Pharmacokinetic Endpoint | 10 |
| 27 | 5.2 | Secondary Pharmacokinetic Endpoints | 11 |
| 28 | 6. MEASI | SUREMENTS AND EVALUATIONS | 11 |
| 29 | 6.1 | Study Data | 11 |
| 30 | 6.2 | Plasma Samples | 11 |
| 31 | 7. SAMPI | PLE SIZE AND ANALYSIS PLAN | 12 |
| 32 | 8.1 | Sample Size | 12 |
| 33 | 8.2 | Statistical and Pharmacokinetic Analysis | 12 |
| 34 | 8. DATA | COLLECTION AND MANAGEMENT PLAN | 12 |
| 35 | 8.1 | Database System Overview | 12 |
| 36 | 8.2 | Case Report Forms and Data Entry | 12 |
| 37 | 9. SAFET | ΓΥ | 12 |
| 38 | 10. REFE | ERENCES | 13 |
| 39 | | | |
| 40 | | | |
| 41<br>42 | | | |
| 43 | | | |
| 7.5 | | | |

#### 1. INTRODUCTION

Peritoneal dialysis (PD) is a form of renal replacement therapy indicated for those with acute kidney injury or end stage renal disease (ESRD). In 2013 PD was utilized in approximately 7% of the 660,000 prevalent patients with ESRD in the United States. Within that time, the prevalence of PD has seen an increase by over 30% between 2007 – 2014.¹ During PD, a hyperosmolar solution is introduced into the peritoneal cavity allowing solute exchange between the dialysate-contained in the cavity and blood from the perfused peritoneum. A concentration gradient is thus created allowing ultrafiltration and diffusional clearance of toxic materials. PD fluids are available as glucose-based or non-glucose based solutions. Commonly prescribed glucose-based PD solutions have been associated with peritoneal membrane injury and negative systemic effects leading to suboptimal patient and technique survival. On the other hand, newer non-glucose based solution marketed in the United States have shown to improve fluid removal during long dialysis exchanges and offer greater peritoneal membrane protection.²

### **Principles of Peritoneal Dialysis**

Currently, two modalities of PD exist and is individualized based on patient and life-style specific factors. Continuous ambulatory peritoneal dialysis (CAPD) allows 4 – 5 exchanges performed manually whereas automated peritoneal dialysis (APD) involves continuous, automated, cyclical exchanges performed by a device at home during the night.<sup>3</sup> APD offers advantages over CAPD by allowing fluid-free or "dry" daytime dwells thereby permitting those who require PD liberty for their activities of daily living. In addition, several other advantages such as lower incidences of infection and hernias, enhanced solute clearances, and positive psychosocial impact have been reported.<sup>3</sup> Overall, the prevalence of APD has been increasing throughout the years as the number of patients utilizing CAPD declines.<sup>4</sup>

#### **Vancomycin in Peritoneal Dialysis**

Peritonitis is a common complication in PD and accounts for a large portion of hospital readmission and mortality.<sup>1,5</sup> In addition, severe or prolonged peritonitis can lead to membrane failure prompting the switch from PD to hemodialysis. The International Society of Peritoneal Dialysis (ISPD) recommends intraperitoneal administration as the preferred route to deliver antibiotics in the absence of systemic bacteremia.<sup>5</sup> Vancomycin is the most common antibiotic recommended and has notable gram-positive coverage used empirically during suspected peritonitis.

#### Rationale for the Proposed Study

Vancomycin is eliminated unchanged in the urine through glomerular filtration and is best characterized by a distribution and elimination phase following parenteral administration. Vancomycin's bactericidal activity is considered time-dependent with the ratio of the 24-hour area-under-the-concentration (AUC) versus time/minimal-inhibitory concentration (MIC) ratio (AUC/MIC) being the best pharmacokinetic/pharmacodynamic predictor of effectiveness. The preferred AUC/MIC ratio is  $\geq$  400. Dosing in the range of 15-30 mg/kg is recommended by several

86

87

88

89 90

91

92

93 94

95

96

97 98

99

100

101

102103

104

105

106

107108

109

110

111112

113114

115

116

117118

119120

121122

123

professional societies including ISPD to maintain a serum concentration level of 15 mg/L in order to maximize efficacy and reduce toxicity, although this trough is only loosely correlated with corresponding AUC/MIC.<sup>5,6</sup> Furthermore, the evidence supporting this recommended trough is essentially nonexistent in PD patients on APD, where data on vancomycin bioavailability and clearance with varying degrees of peritoneal function is sparse. In addition, early pharmacokinetic studies were conducted only in patients on CAPD modalities, glucose-based prescriptions, or those on intravenous vancomycin.<sup>7-9</sup> Lastly, the relationship between serum concentration and site of action at the peritoneal cavity wall is not established. In totality, the goal is to close the knowledge gap in this very common use of vancomycin.

Although the ISPD advisory committee on peritonitis management recommends a 25% increase in antibiotic dose in non-anuric patients, residual kidney function may affect the exposure, clearance, distribution and serum half-life for those antibiotics administered. This however is an empiric recommendation and there is no formal quantification of how residual kidney function (RKF) may impact pharmacokinetics. The impact on RKF on vancomycin in PD is also lacking. RKF is critical for the welfare and survival of PD patients. Indeed, 2 large multicenter studies, the Netherlands Cooperative Study on the Adequacy of Dialysis (NECOSAD-2) (AJKD;41:1293-2302, 2003) and the Canada/USA Peritoneal Adequacy Study (CANUSA) (JASN, 12:2158-2162, 2001), both have shown statistically significant (by multivariable analyses) 12% reductions in mortality per ml/min/1.73 m<sup>2</sup> residual GFR increase or per 5L/week residual GFR increase, respectively. Hence, it is important to assess vancomycin pharmacokinetics in PD patients with RKF for two reasons. First, the enhanced vancomycin clearance of RKF may result in under-dosing and secondly, overdosing may result in nephrotoxicity and loss of critically important RKF. This presents a challenge when considering the bi-exponential pharmacokinetic behavior of vancomycin and produces a significant source of variability allowing controversy in the role of monitoring serum vancomycin in patients on APD. 10,11

Interestingly, a recent retrospective analysis examining residual renal function and peritonitis outcomes show that the odds of peritonitis treatment failure for those with urinary creatinine clearances of greater than 5 mL/min were greater when compared to those who were anuric.<sup>12</sup> These associations further challenge the need for optimal vancomycin dosing strategies in patients on rapid-cycling modalities to maximize the efficacy, safety, and cost.

Moreover, icodextrin a non-glucose based PD fluid, is an increasingly used PD dialysate solution to complement conventional glucose-based PD fluids. Commonly prescribed glucose-based PD solutions have been associated with peritoneal membrane injury and negative systemic effects leading to suboptimal patient and technique survival. Non-glucose based solutions such as icodextrin marketed in the United States have shown to improve fluid removal during long dialysis exchanges and offer greater peritoneal membrane protection. In-vitro studies conducted with 7.5% icodextrin demonstrate physical compatibility and chemical stability, however there is a lack of information for the clearance, stability and effect on the minimum inhibitory

#### **PROTOCOL**

129

140141

142

143

144

- 124 concentration of vancomycin in-vivo. 13 As there will be increasing use of icodextrin,
- characterization of vancomycin pharmacokinetics will be important.
- Therefore, this current study aims to explore the pharmacokinetics and pharmacodynamics of
- intraperitoneal administered vancomycin in un-infected subjects on APD and explore the in-vivo
- behavior of vancomycin in 7.5% icodextrin PD solution.

#### 2. STUDY OBJECTIVES

#### 130 2.1 Primary Objective

- Characterize the pharmacokinetic profile of vancomycin in serum, urine, and dialysate following a single intermittent intraperitoneal dose of vancomycin in non-infected
- patients on automated peritoneal dialysis

#### 134 2.2 Secondary Objectives

- Examine the relationship between residual kidney function and vancomycin clearance using serum, dialysate and urine
- Describe the safety, tolerability, and stability of intraperitoneal vancomycin when administered in a 7.5% icodextrin-containing dialysis solution

#### 2.3 Exploratory Objectives

- Investigate dosing recommendations and adjustments based on population pharmacokinetic parameters generated from serum and dialysate concentrations in adult patients on APD
- Correlate the peritoneal transport function, measured using the peritoneal equilibration test (PET), to vancomycin pharmacokinetics
- Correlate dialysis adequacy, measured as a function of peritoneum urea clearance, time, and volume of dialyzer fluid (Kt/V), to vancomycin pharmacokinetics

#### 3. STUDY DESIGN

#### 148 3.1 Overview and Design

- 149 This is a prospective, single-site, open-label, pharmacokinetic study of vancomycin in infection-
- 150 negative healthy adult patients on peritoneal dialysis. Prospective patients will be identified
- through Thomas Jefferson University Hospital nephrology practice. Subjects will be asked to
- consent prior to participation in the study. The majority of research activities will take place at
- the Thomas Jefferson University Clinical Research Unit (CRU).
- Subjects will be on an APD regimen consisting of a 12-hour overnight dwell followed by a 9-hour
- on-cycler exchange (figure 1). Vancomycin will be administered via intraperitoneal injection in 1
- liter of icodextrin solution. There will be 4 exchanges during the 9-hour exchange period. A sparse
- sampling approach will be used in collecting blood samples. A total of 16 blood samples will be
- 159 collected.

160 161



**Figure 1.** Schematic depiction of APD regimen.

206

207

#### Schedule & Procedures

A schematic is illustrated in figure 2 and study procedure detailed in table 1.



Figure 2. Study day and sampling schematic

| Procedures | | Screening<br>(Day -30) | Pre-study Day<br>(Day - 1) | Study<br>Day 1 | Study<br>Day 2 | Study<br>Day 3 | Study<br>Day 4 | Study<br>Day S | Study<br>Day 6 | Study<br>Day 7 | Post-study<br>Rollow-up (+7*<br>to 10 days) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| As | ssessment of Eligibility | x | | | | | | | | | |
| | Signed Consent Form | x | | | | | | | | | |
| | Medical History | x | | | | | | | | | |
| Conco | mitant Medication Review | x | × | x | × | × | × | × | x | × | |
| | Pregnancy Test | × | | | | | | | | | _ |
| = | Complete Blood Count | x | | | | | | | | | <b>x</b> <sup>5</sup> |
| Clinical Laboratory | Comprehensive Metabolic<br>Panel | x | | x <sup>4</sup> | x <sup>4</sup> | x <sup>4</sup> | x <sup>4</sup> | x <sup>4</sup> | x <sup>4</sup> | x <sup>4</sup> | x <sup>5</sup> |
| 5 | HIV, Hepatitis B & C | X1 | | | | | | | | | |
| Ü | Alcohol & Drug Screen | x | | | 7 | | | | | | |
| | Urinary Creatinine & Urea | | | x | × | x | × | × | x | x | |
| S S | Physical Exam | x | | x | × | × | × | × | x | × | x |
| 200 | Vital Signs | x | | x | × | x | х | x | x | x | x |
| Clinical Procedures | Electrocardiogram | x | | | | | | | | | |
| tory | PK Blood Sample | | | x | x | х | x | x | x | х | |
| Research Laboratory | PK Urine Sample | | | x | x | x | x | x | x | x | |
| Resear | PK Dialysate Sample | | | × | x | x | x | x | x | x | |
| Treatment | Vancomycin 20 mg/kg | | | x² | | | | | | | |
| Asses | Assessment of Adverse Events | | | × | × | x | × | × | x | x | × |
| CI | RU Evening Admission | | × | | | | | | | | |
| | CRU Discharge | | | x³ | | | | | | | |

<sup>&</sup>lt;sup>1</sup> HIV/HBV/HCV information will be obtained from previous medical history. If the information is not available or a test was performed for  $\geq$  2 months, then a test will be performed during pre-screening.

**Table 1.** Summary of study procedures from pre-study to post-study follow-up.

<sup>&</sup>lt;sup>2</sup> Vancomycin is dosed intraperitoneally in 1-liter of 7.5% icodextrin solution.

<sup>&</sup>lt;sup>3</sup> Subjects are ambulatory after study day 1.

<sup>&</sup>lt;sup>4</sup> Subjects will have serum creatinine analyzed within the PK sample.

<sup>&</sup>lt;sup>5</sup> Laboratory assessments will be ordered at the discretion of the physician-investigator.

<sup>&</sup>lt;sup>6</sup> If patient cannot produce urine, a urine drug screen will not be performed.

<sup>&</sup>lt;sup>7</sup> If patient cannot produce urine, urinary creatinine and urea will not be performed.

#### 297 Screening Visit for All Subjects (Day -30)

- Subjects will be screened up to approximately 30 days prior to beginning the study. The screening visit will consist of:
- 300 Previous medical history
  - HIV
  - Hepatitis B
  - Hepatitis C
  - Alcohol and drug screen
    - If the patient cannot produce urine, then a urine drug screen will not be performed and should not be considered a protocol deviation or exclusionary of participation in study
- 308 Physical examination
- 309 Patient consent
- 310 Vital signs

301 302

303

304

305

306 307

320 321

322

323

324 325

326

327328

329

330

331

332333

334

335

336

337

- 311 Electrocardiogram (ECG)
- 312 Complete blood count
- 313 Comprehensive metabolic panel

#### 314 Study Days -1 - 1

- 315 Physical exam and vital signs
- 316 Urine will be immediately voided prior to dosing
- Administer vancomycin 20 mg/kg in 1 liter of 7.5% icodextrin intraperitoneally over
   approximately 10 to 15 minutes
- 319 Off-Cycler Schedule (12 hours)
  - Blood samples will be obtained during the first 12-hour overnight dwell. A total of two samples will be taken between the time interval following dosing up until hour 12
  - Vancomycin and serum creatinine will be evaluated from blood samples collected
  - Dialysate samples will be obtained during the first 12-hour overnight dwell. A total of two samples will be taken between the time interval following dosing up until hour
     12
  - o Any urine voided will be collected between the time following dosing up until hour 12
    - If the patient cannot produce urine, then a urine sample will not be possible and should not be considered a protocol deviation

#### On-Cycler Schedule (9 hours)

- Blood will be sampled prior to and after each exchange. Since there are four exchanges, it is anticipated that a total of 8 samples will be obtained during the 9hour on-cycler exchange period
- Vancomycin and serum creatinine will be evaluated from blood samples collected
- Wasted dialysate from each exchange will be collected and stored
  - Urine will be collected and pooled
    - If the patient cannot produce urine, then a urine sample will not be possible and should not be considered a protocol deviation
- 338 Discharge from CRU

#### 339 **Study Days 2 – 7**

340

341

342343

344

345

346

347

348

349 350

351

357

358

359

362

363

364

366

367

- An additional 6 blood samples will be taken following study day 1, totaling 1 sample per day for the days the patient can come in. A minimum of 4 samples must be collected. If a patient cannot come in for at least 4 of the six days or blood cannot be obtained, it will be considered a protocol deviation. This will be done ideally in the morning, but at a time that takes into consideration subject availability and scheduling
- Vancomycin and serum creatinine will be evaluated from blood samples collected
- Vital signs will be taken
  - Ambulatory dialysate and 24-hour urine will be collected from the subjects
    - If the patient cannot produce urine, then a urine sample will not be possible and should not be considered a protocol deviation

#### Post-study follow up

The post study visit will include post-study labs (at the investigator or co-investigator's discretion)\*, physical exam, vital signs, and adverse event assessment obtained from the end of study. \* As peritoneal dialysis patients come in to clinic regularly and have routine standard of care labs drawn, these may be used to evaluate follow- up safety as long as they are scheduled to be drawn no later than 17 days post dose.

#### 4. STUDY POPULATION

#### 4.1 Inclusion Criteria

- Adult male or females between 18 85 years old
- On a PD regimen for > 3 months prior to study initiation

#### 361 4.2 Exclusion Criteria

- Clinically significant disease unrelated to renal impairment or deemed unfit by the investigator
- Allergy or hypersensitivity to vancomycin or icodextrin-containing dialysis solution
- 365 Active peritonitis infection
  - Hospitalization within < 3 months</p>
    - Previous intraperitoneal antibiotic treatment within 2 months
- Previous intravenous vancomycin treatment within 2 months
- 369 Hemoglobin < 9 g/dL
- 370 Pregnant or breast-feeding women

#### 371 5. STUDY ENDPOINTS

#### 372 5.1 Primary Pharmacokinetic Endpoint

- 373 Pharmacokinetic parameters such as the maximum serum concentration (C<sub>max</sub>), time to
- maximum concentration ( $T_{max}$ ), area under the concentration-time curve (AUC), half-life ( $t_{1/2}$ ),
- volume of distribution (VD), dialysate and systemic clearance, and inter-subject variability of
- vancomycin in subjects on APD will be estimated following a non-compartmental analysis (NCA).

| | Pharmacokinetics of Vancomycin in Automated Peritoneal Dialysis PROTOCOL |
|---|---|
| 377<br>378<br>379 | Dialysate parameters will be estimated following an NCA analysis. Systemic bioavailability from the peritoneal cavity and absorption constant will be estimated. |
| 380<br>381<br>382<br>383<br>384<br>385 | 5.2 Secondary Pharmacokinetic Endpoints Residual kidney function as it relates to vancomycin will be assessed based on vancomycin total urinary clearance and cumulative drug excretion. The total dialysate clearance of vancomycin will be explored based on the biological fluids obtained. The safety, tolerability, and stability of vancomycin in 7.5% icodextrin solution will also be described. |
| 386<br>387<br>388<br>389<br>390 | 5.3 Exploratory Pharmacokinetic-Pharmacodynamic Endpoints Parameters generated from the non-compartmental analysis will be used to parameterize the population pharmacokinetic model to explore various dosing profiles. The AUC/MIC ratio will be explored to correlate exposures to the effect of vancomycin in patients on APD. |
| 391<br>392 | 6. MEASUREMENTS AND EVALUATIONS 6.1 Study Data |
| 392<br>393<br>394 | Patient data will be recorded in a secured study database. Elements of interest to the study include: |
| 395<br>396<br>397<br>398<br>399<br>400<br>401<br>402<br>403<br>404<br>405<br>406<br>407 | <ul> <li>Patient demographics <ul> <li>Age</li> <li>Sex</li> <li>Height</li> <li>Weight</li> <li>Race</li> <li>Cause of ESRD</li> </ul> </li> <li>Laboratory parameters <ul> <li>Serum creatinine (SCr)</li> <li>Urinary creatinine</li> <li>Blood Urea Nitrogen (BUN)</li> <li>Urine urea</li> <li>Liver function</li> </ul> </li> </ul> |
| 408<br>409 | 6.2 Plasma Samples Samples will be processed per laboratory protocol in the laboratory manual. |

6.3

6.4

410

411

412

413

**Dialysate Samples** 

**Urine Samples** 

Samples will be processed per laboratory protocol.

Samples will be processed per laboratory protocol.

Page **11** of **14** 

### 414 7. SAMPLE SIZE AND ANALYSIS PLAN

- 415 8.1 Sample Size
- Due to the exploratory nature of this pharmacokinetic study, no formal sample size calculation
- was performed. A total of 4 subjects will be enrolled.
- 418 8.2 Statistical and Pharmacokinetic Analysis
- 419 A non-compartmental analysis (NCA) will be utilized to estimate vancomycin pharmacokinetic
- parameters in patients on APD. The values generated from the NCA will be used to parameterize
- 421 the population pharmacokinetic model.

422

- Data from all patients will be analyzed simultaneously using nonlinear mixed-effects modelling
- 424 software (NONMEM). A base model will be developed to characterize the data. Covariate analysis
- will also be evaluated in the model to explain for any intra- and inter-patient PK variability. Model
- 426 qualification will be validated by using appropriate internal validation procedures based on the
- data and model development process.

### 428 8. DATA COLLECTION AND MANAGEMENT PLAN

- 429 8.1 Database System Overview
- Data will be recorded and accessed using Research Electronic Data Capture, known as REDCap.
- 431 REDCap is a secure web application designed for building and managing database information
- 432 and meets compliance standards mandated by the Health Insurance Portability and
- 433 Accountability Act (HIPAA) and FDA 21 CFR Part 11. Data files can be conveniently exported into
- various data formats (e.g. Microsoft Excel, SAS Statistical Software, R, SPSS, or STATA) for further
- 435 analysis.
- 436 8.2 Case Report Forms and Data Entry
- 437 Clinical and demographic data will be collected from paper source documents. Information will
- 438 be entered into an electronic case report form (eCRF). Each enrolled subject's eCRF will then be
- 439 transcribed into REDCap and will serve as a central repository of all enrolled subjects in the study.
- 440 A data monitor will monitor the accuracy of the study charts and data entry.
- 441 8.3 Case Report Form Storage and Backup
- The eCRF will be stored in the Department of Pharmacology & Experimental Therapeutics
- secured server. Access will only be granted by the principal investigator or co-investigators.
- 444 9. SAFETY
- Vancomycin has been previously studied in non-infected patients on peritoneal dialysis. In
- addition, the dose selected in this study is not devoid of the doses used in previous studies
- administered intravenously or through the intraperitoneal route.<sup>7,9</sup> The safety and tolerability of
- vancomycin administered through the intraperitoneal route will be assessed in this study by
- description of vital signs, physical examinations, and laboratory safety evaluations. In
- 450 addition, continual serum concentration monitoring through blood sampling will be performed

as part of this research study. In addition, the likelihood for rare adverse events to vancomycin 451 452 such as ototoxicity will be unlikely to occur based on the minimal dose used compared to 453 literature. 14 Nephrotoxicity from a single IP 20 mg/kg dose of vancomycin would be extremely 454 unlikely in stable, non-septic patients receiving no other potentially nephrotoxic medications or 455 intravenous contrast. Major risk factors for nephrotoxicity related to vancomycin dosing include large daily doses (> 4grams/day), prolonged duration, and concurrent potentially toxic antibiotics 456 457 (aminoglycosides or piperacillin-tazobactam), none of which apply to this study protocol. Other associated adverse events relating to vancomycin such as anaphylaxis and development of 458 Clostridium difficile infections are considered unlikely. 15 In the event that greater than two 459 unexpected and treatment related serious adverse events occur, the study will be halted until 460 461 review from an independent study monitor is conducted. Cumulative blood draws will be 462 restricted to less than 3 mL per sampling procedure and will be kept in strict accordance with 45 463 CFR 46.402(a) OHRP expedited review categories. Subjects who enrolled in the study will already 464 have hemoglobin levels greater than 9 g/dL eliminating the concern for anemia requiring blood 465 transfusion.

#### 10. REFERENCES

- 1. Chan L, Poojary P, Saha A, et al. Reasons for admission and predictors of national 30-day readmission rates in patients with end-stage renal disease on peritoneal dialysis. *Clin Kidney J.* 2017;10(4):552-559.
- 470 2. Garcia-Lopez E, Lindholm B, Davies S. An update on peritoneal dialysis solutions. *Nat Rev* 471 *Nephrol.* 2012;8(4):224-233.
- 472 3. Rabindranath KS, Adams J, Ali TZ, Daly C, Vale L, Macleod AM. Automated vs continuous 473 ambulatory peritoneal dialysis: a systematic review of randomized controlled trials. *Nephrol Dial* 474 *Transplant*. 2007;22(10):2991-2998.
- 475 4. Manley HJ, Bailie GR. Treatment of peritonitis in APD: pharmacokinetic principles. *Semin Dial.* 476 2002;15(6):418-421.
- Li PK, Szeto CC, Piraino B, et al. ISPD Peritonitis Recommendations: 2016 Update on Prevention and Treatment. *Perit Dial Int.* 2016;36(5):481-508.
- 479 6. Rybak M, Lomaestro B, Rotschafer JC, et al. Therapeutic monitoring of vancomycin in adult
  480 patients: a consensus review of the American Society of Health-System Pharmacists, the
  481 Infectious Diseases Society of America, and the Society of Infectious Diseases Pharmacists. *Am J*482 *Health Syst Pharm.* 2009;66(1):82-98.
- Morse GD, Farolino DF, Apicella MA, Walshe JJ. Comparative study of intraperitoneal and intravenous vancomycin pharmacokinetics during continuous ambulatory peritoneal dialysis.
   Antimicrob Agents Chemother. 1987;31(2):173-177.
- 8. Bunke CM, Aronoff GR, Brier ME, Sloan RS, Luft FC. Vancomycin kinetics during continuous ambulatory peritoneal dialysis. *Clin Pharmacol Ther*. 1983;34(5):631-637.
- 488 9. Manley HJ, Bailie GR, Frye RF, McGoldrick MD. Intravenous vancomycin pharmacokinetics in automated peritoneal dialysis patients. *Perit Dial Int.* 2001;21(4):378-385.
- 490 10. Fish R, Nipah R, Jones C, Finney H, Fan SL. Intraperitoneal vancomycin concentrations during 491 peritoneal dialysis-associated peritonitis: correlation with serum levels. *Perit Dial Int.* 492 2012;32(3):332-338.
- 493 11. Stevenson S, Tang W, Cho Y, et al. The role of monitoring vancomycin levels in patients with peritoneal dialysis-associated peritonitis. *Perit Dial Int.* 2015;35(2):222-228.

- Whitty R, Bargman JM, Kiss A, Dresser L, Lui P. Residual Kidney Function and Peritoneal Dialysis-Associated Peritonitis Treatment Outcomes. *Clin J Am Soc Nephrol.* 2017;12(12):2016-2022.
- 497 13. Ranganathan D, Naicker S, Wallis SC, Lipman J, Ratanjee SK, Roberts JA. Stability of Antibiotics 498 for Intraperitoneal Administration in Extraneal 7.5% Icodextrin Peritoneal Dialysis Bags (STAB 499 Study). *Perit Dial Int.* 2016;36(4):421-426.
- Tokgoz B, Somdas MA, Ucar C, et al. Correlation between hearing loss and peritonitis frequency
   and administration of ototoxic intraperitoneal antibiotics in patients with CAPD. *Ren Fail.* 2010;32(2):179-184.
- 503 15. Sun Y, Huskey RL, Tang L, et al. Adverse effects of intravenous vancomycin-based prophylaxis during therapy for pediatric acute myeloid leukemia. *Antimicrob Agents Chemother*. 2017.